CLINICAL TRIAL: NCT00905957
Title: Transversus Abdominis Plane Block For Renal Transplant Recipients: A Randomized Controlled Double-blinded Study
Brief Title: Transversus Abdominis Plane Block For Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: KARIM MUKHTAR, ROYAL LIVERPOOL AND BROADGREEN UNIVERSITY HOSPITALS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3818
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2010-10

CONDITIONS: Disorder Related to Renal Transplantation; Pain
Keywords: transversus abdominis plane block; relief
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus abdominis plane (TAP) Group (Active Comparator): Patients will receive a TAP block using a local anaesthetic agent after induction of anaesthesia
  Interventions: Procedure: TAP block
- Control Group (Placebo Comparator): Patients will receive a TAP block using a placebo after induction of anaesthesia
  Interventions: Procedure: TAP block with placebo

INTERVENTIONS:
Procedure: TAP block — TAP block using 20 ml of a local anaesthetic agent will be used in the treatment group
  Arms: Transversus abdominis plane (TAP) Group
Procedure: TAP block with placebo — TAP block using a placebo after induction of anaesthesia
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of a local anaesthetic injection in the plane between the abdominal muscles in reducing the amount of pain relief required after surgery.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of transversus abdominis plane block in reducing the morphine requirements after renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant recipients
* 18 to 75 years

Exclusion Criteria:

* allergy to local anaesthetics
* chronic pain
* refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in first 24 hours after renal transplantation | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Liverpool and Broadgreen University Hospitals, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] Gulyam Kuruba SM, Mukhtar K, Singh SK. A randomised controlled trial of ultrasound-guided transversus abdominis plane block for renal transplantation. Anaesthesia. 2014 Nov;69(11):1222-6. doi: 10.1111/anae.12704. Epub 2014 Jun 28. PMID 24974901